CLINICAL TRIAL: NCT05605262
Title: Effects of 100% Medical Grade Manuka Honey on Re-epithelialization Post Tympanoplasty in the Case of Mucosal Type Chronic Suppurative Otitis Media (CSOM) - A Prospective Double-blinded Randomized Controlled Trial
Brief Title: Effects of 100% Medical Grade Manuka Honey on Tympanic Membrane Reconstruction Healing.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21040425
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Otitis Media, Suppurative; Tympanic Membrane Perforation
Keywords: Chronic Suppurative Otitis Media; Manuka Honey; Wound Healing; Re-epithelialization; Tympanoplasty; Tympanic Membrane
MeSH Terms: conditions — Otitis Media, Suppurative; Tympanic Membrane Perforation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Manukamed - 100% sterile manuka honey
  Interventions: Drug: Manukamed - Manukapli 100% sterile honey wound dressing - Premium medical grade 16+ Leptospermum Scoparium New Zealand honey
- Control (No Intervention): No intervention was given. Participants receive standard wound care of the tympanic membrane which includes 0.3% Ofloxacin otic ear drops which were used twice a day for 5 days.

INTERVENTIONS:
Drug: Manukamed - Manukapli 100% sterile honey wound dressing - Premium medical grade 16+ Leptospermum Scoparium New Zealand honey — After surgical reconstruction of the tympanic membrane by grafting, Manukamed - Manukapli 100% Sterile honey wound dressing is applied onto the gelfoam to close the area, followed by an antibiotic tampon.
  Other Names: Manukamed - Manukapli 100% sterile honey wound dressing
  Arms: Intervention

SUMMARY:
Throughout history, honey has been recognized for its healing properties. The use of honey for its medicinal properties dates back to 2200 BCE.

The purpose of this clinical trial is to learn about the healing effects of 100% medical grade Manuka honey in participants with Chronic Suppurative Otitis Media of the mucosal type.

The main question it aims to answer is: Can 100% Manuka honey given at the time of Tympanoplasty improve the re-epithelialization (healing process) of the tympanic membrane compared to controls?

Participants in the intervention group will receive a wound dressing of 100% medical grade Manuka honey after reconstructive surgery of the tympanic membrane.

Researchers will compare the intervention group to the control group to see healing process.

DETAILED DESCRIPTION:
The aim of the present study is to conduct a randomized clinical trial to compare the effect of 100% sterile Manuka honey on re-epithelialization of the tympanic membrane post Tympanoplasty compared to the control group. The investigation will involve 64 participants with Chronic Suppurative Otitis Media of the mucosal type, who will be randomly put into two groups (intervention or control), where the intervention group will receive a dressing of 100% sterile Manuka honey during surgery. Results of this study will inform practitioners as to the potential benefits of 100% sterile Manuka honey on the re-epithelialization of the tympanic membrane.

ELIGIBILITY:
Inclusion Criteria:

* Participants of 18 - 45 years of age.
* Participants with Chronic Suppurative Otitis Media of the mucosal type.
* Provision of signed and dated informed consent form. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Participants who previously received surgical therapy for Chronic Suppurative Otitis Media or have recurrent or residual disease.
* Participants with anatomical pathology results showing and/or suspecting a tumor.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-06-13 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Weekly Evaluation of Tympanic Membrane Re-epithelialization Post-tympanoplasty | 2 weeks (14 days following surgery)
  Epithelialization of the tympanic membrane was measured using an indicator tool utilizing a filter paper (5 mm in width and 10 mm in length) with a water-based ink on one end as the indicator. Exposure of the indicator to the exudate on the surface of the tympanic membrane will reveal the status of the wound (wet/ dry).

SECONDARY OUTCOMES:
Weekly Evaluation of Tympanic Membrane Re-epithelialization Post-tympanoplasty | 3 weeks (21 days following surgery)
  Epithelialization of the tympanic membrane was measured using an indicator tool utilizing a filter paper (5 mm in width and 10 mm in length) with a water-based ink on one end as the indicator. Exposure of the indicator to the exudate on the surface of the tympanic membrane will reveal the status of the wound (wet/ dry).
Weekly Evaluation of Tympanic Membrane Re-epithelialization Post-tympanoplasty | 4 weeks (28 days following surgery)
  Epithelialization of the tympanic membrane was measured using an indicator tool utilizing a filter paper (5 mm in width and 10 mm in length) with a water-based ink on one end as the indicator. Exposure of the indicator to the exudate on the surface of the tympanic membrane will reveal the status of the wound (wet/ dry).
Weekly Evaluation of Tympanic Membrane Re-epithelialization Post-tympanoplasty | 5 weeks (35 days following surgery)
  Epithelialization of the tympanic membrane was measured using an indicator tool utilizing a filter paper (5 mm in width and 10 mm in length) with a water-based ink on one end as the indicator. Exposure of the indicator to the exudate on the surface of the tympanic membrane will reveal the status of the wound (wet/ dry).
Weekly Evaluation of Tympanic Membrane Re-epithelialization Post-tympanoplasty | 6 weeks (42 days following surgery)
  Epithelialization of the tympanic membrane was measured using an indicator tool utilizing a filter paper (5 mm in width and 10 mm in length) with a water-based ink on one end as the indicator. Exposure of the indicator to the exudate on the surface of the tympanic membrane will reveal the status of the wound (wet/ dry).
Evaluation of Ototoxicity | 5 weeks (35 days following surgery)
  Hearing function will be evaluated by conducting a Brain Evoked Response Audiometry exam. If the BERA results show decreased stimulus of more than 10 decibels, treatment for sudden deafness is started immediately.

CONTACTS AND LOCATIONS:
Overall Officials: Harim Priyono, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Faculty of Medicine - University of Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
If requested, data records without identifying patient information can be shared

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT05605262/Prot_SAP_000.pdf